CLINICAL TRIAL: NCT02116400
Title: Neuropsychological Characterization of Patients With Bipolar Disorder and a History of Suicide Attempt
Acronym: DECISIDAIRE
Status: Withdrawn | Type: Observational
Why Stopped: The primary investigator moved.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2012/FC-02; 2012-A01673-40 (Other: RCB number)
Record Dates: First submitted 2014-04-15; First posted 2014-04-16 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Bipolar Disorder
Keywords: Suicidal ideation
MeSH Terms: conditions — Bipolar Disorder; Suicidal Ideation | interventions — Interviews as Topic; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Leftover serum samples will be stored in the Nîmes University Hospital Biothèque.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Suicidal: Patients in this group have had suicidal behaviour according to the C-SSRS score.
  Intervention: Interview Intervention: Neuropsychological testing Intervention: Serum concentration of lithium or sodium divalproate.
  Interventions: Other: Interview; Other: Neuropsychological testing; Biological: Serum concentration of lithium or sodium divalproate.
- Not suicidal: Patients in this group have not had suicidal behaviour according to the C-SSRS score.
  Intervention: Interview Intervention: Neuropsychological testing Intervention: Serum concentration of lithium or sodium divalproate.
  Interventions: Other: Interview; Other: Neuropsychological testing; Biological: Serum concentration of lithium or sodium divalproate.

INTERVENTIONS:
Other: Interview — All patients are interviewed at the BEC. Questionnaires and scores are administered. See endpoints.
Other: Neuropsychological testing — Neuropsychological tests are administered (requires computer use). See endpoints.
Biological: Serum concentration of lithium or sodium divalproate. — Venous blood is drawn and tested for serum concentration of lithium or sodium divalproate.

SUMMARY:
The main objective of this study is to evaluate decision-making using the Iowa Gambling Task (IGT) among patients with euthymic bipolar disorder according to their personal history of suicide attempt ("suicidal" vs. "not suicidal ").

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. Evaluate other aspects of cognitive functioning (using the Tower of London, the Probabilistic Reversal-learning task, the Rey Complex Figure, the Reading the Mind in the Eyes test) in euthymic patients with bipolar disorder, depending on the presence or absence of a history of suicide attempt; B. Explore performance on neuropsychological tests depending on the type of therapy administered (lithium salts or valproate monotherapy or in combination with other mood stabilizers); C. Explore a possible relationship between circulating levels of lithium or sodium divalproex results and different neuropsychological tests; D. Establishment of a biobank for this population with leftover blood samples following serum lithium or divalproex testing.

ELIGIBILITY:
Inclusion Criteria:

* The patient was correctly informed about the study
* The patient must be insured or beneficiary of a health insurance plan
* The diagnosis of bipolar disorder is confirmed by the doctor referring the patient to the BEC and confirmed during the preliminary interview at the BEC
* The patient is euthymic on the day of inclusion. This is supported by a short psychiatric interview conducted at the BEC and the completion of the depression and mania scales (score <= 7 on the HDRS questionnaire and score <= 7 on the YMRS questionnaire).
* The patient is prescribed a mood stabilizer based on lithium or divalproex.

Exclusion Criteria:

* The patient is under judicial protection, under tutorship or curatorship
* The patient formalizes his/her opposition to the studyd
* It is impossible to correctly inform the patient
* The patient has mental retardation
* The patient has practiced substance abuse or dependence within the 6 months prior to study inclusion (alcool, cannabis, opiates, psychostimulants)
* The patient does not meet euthymic criteria (score <= 7 on the HDRS questionnaire and score <= 7 on the YMRS questionnaire).

Uninclusion Criteria:

* The patients withdraws consent during the study
* The patient does not understand directions necessary for the neurpsychological tasks
* The patient is not able to use a computer to complete the neuropsychological tasks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients are recruited via the Bipolar Expert Centres (BEC) at the participating hospitals. Euthymic bipolar patients requiring a lithium or divalproex -based mood stabilizer will be included.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline (day 0)
The Iowa Gambling Task | Baseline (day 0)

SECONDARY OUTCOMES:
The Tower of London Test | Baseline (day 0)
The Probabilistic Reversal Learning Task | Baseline (day 0)
The Rey Osterreith Complex Figure Task | Baseline (day 0)
The Baron-Cohen Test | Baseline (day 0)
Serum concentration for divalproate (mg/l) | Baseline (day 0)
Serum concentration for lithium (mEq/l) | Baseline (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Cyprien, MD, Principal Investigator — CHRU de Nîmes - Hôpital Universitaire Carémeau